CLINICAL TRIAL: NCT07332897
Title: Motor Relearning Program Combined With Neck Stabilization Exercises in Subacute Stroke
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Stroke (Subacute)
Keywords: Motor relearning program, neck stabilization exercises, stroke (subacute)
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nterventional Group A (Experimental): Experimental: Interventional Group A
  These patients will be treated by neck stabilization exercises and motor relearning program with 3 sets of 10 repetitions each and 10 seconds along with 10 successful attempts in one session. Delivered five times a week for four weeks For this, participants will be given a comfortable assisted sitting and transition to standing position.
  Interventions: Other: Motor relearning program combined with neck stabilization exercises
- Interventional Group B (Active Comparator): Active Comparator: Interventional Group B
  These patients will be treated by routine physical therapy exercises with motor relearning program with three sets of 10 repetitions each, squeeze hold for 10 seconds, stretch hold for 30 seconds repetitions in one session for 4 weeks, five times every week. For this, participants will be given a comfortable supine lying transition to assisted sitting position.
  Interventions: Other: Motor relearning program combined with routine physical therapy

INTERVENTIONS:
Other: Motor relearning program combined with neck stabilization exercises — Neck stabilization exercises and Motor relearning program based functional activities will be performed
  Arms: nterventional Group A
Other: Motor relearning program combined with routine physical therapy — Routine Physical therapy exercises and Motor relearning program based functional activities will be performed
  Arms: Interventional Group B

SUMMARY:
Stroke is a neurological event that leads to significant motor and functional impairments due to disruption of cerebral blood flow. The subacute phase, typically ranging from day of attack up to three months post-stroke, is a critical window for neuroplasticity and functional recovery. The proposed study will find out the effects of motor relearning program combined with neck stabilization exercises for health-related quality of life, sensorimotor function and upper extremity functionality.

DETAILED DESCRIPTION:
This is a randomized clinical trial. Target population is patients suffering from subacute stroke with an MMSE score of 24 and above. Data will be collected from The University of Lahore teaching Hospital and Shadman Medical Center. This study will include 96 participants with 10% dropout ratio, according to the selection criteria. The participants will be randomly divided into two groups through a computer-generated random number table.

Group A will recruit 48 patients to fulfil the inclusion criteria. These patients will undergo a 60 minutes session delivered for four weeks with 5 sessions every week, including warm-up, neck stabilization exercises, cranio-cervical flexion, cervical isometrics, 3 sets x 10 repetitions each 10 seconds hold, eye head coordination drills, 3 sets 60 seconds, focusing on target (right, left, up, down) neck control while reaching, 10 successful attempts, all performed in assisted sitting position. Combined with motor relearning program activities assisted supported sitting & standing grasping and releasing cylinder progressing to cloth, reaching targets forward and sideways, picking objects and transferring over shelves 2 meters apart, Coin stacking, assisted grooming and ADLs (combing hair, turning keys, drinking water) 10 successful attempts of each activity. Group B will recruit 48 patients which fulfill the inclusion criteria. These patients will be treated by routine physical therapy, evidence-based exercises including AAROM of shoulder, elbow & wrist joint, Scapular retraction, Shoulder and elbow isometrics, stretching of pectoralis minor and shoulder internal rotators, therapist assisted PNF diagonals for upper limb (Three sets of 10 repetitions each, squeeze hold for 10 seconds, stretch hold for 30 seconds and motor relearning program activities same as Group A, delivered under supervision over a timeframe of 60 minutes per session for four weeks, 5 times per week. The Statistical analysis will be performed through SPSS Software 21

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed for stroke in subacute phase by a neurologist
* Patients with Mini Mental State Examination score of 24 and above

Exclusion Criteria:

* Patients with accompanying mental Disorders (unable to cooperate)
* Fracture of upper limb in last 6 months
* Recent surgery of upper periphery effecting mobility and motor functionality
* Non consenting to intervention

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Sensorimotor Function | Four weeks
  Sensorimotor function will be assessed by using Urdu translated version of Fugl-Meyer Assessment (FMA) for Upper Extremity (UE)
Upper Limb Functionality | Four weeks
  Functionality, assessed by using Wolf Motor Functional Test
Health Related Quality of Life | Four weeks
  Health Related Quality of life will be assessed by using Stroke Impact Scale

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Shadman Medical Center, Lahore, Punjab Province
  - The University of Lahore Teaching Hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: Undecided